CLINICAL TRIAL: NCT04410835
Title: Psychological Impact and Effect of the Corona Virus (SARS-CoV-2) and COVID-19 Pandemic in Individuals With Psychiatric Disorders - an Online Survey
Brief Title: Psychological Impact of the Corona Virus (SARS-CoV-2) and COVID-19 Pandemic in Individuals With Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 32-363 ex 19/20
Record Dates: First submitted 2020-05-14; First posted 2020-06-01 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Corona Virus Infection; Psychiatric Disorder; Psychological Distress
MeSH Terms: conditions — Coronavirus Infections; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psychiatric patients: Psychiatric patients with ICD-10 (International Statistical Classification of Diseases and Related Health Problems) F2/F3/F4 diagnosis
  Interventions: Diagnostic Test: Online Survey
- Healthy Controls: Participants who do not have a psychiatric disorder or a first degree relative with psychiatric disorder.
  Interventions: Diagnostic Test: Online Survey

INTERVENTIONS:
Diagnostic Test: Online Survey — Psychological questionnaires

SUMMARY:
The aim of this study is to measure current affective symptoms and psychological distress in individuals with severe mental illness during the COVID-19 pandemic using an online questionnaire survey. In addition, this study aims at identifying individual beliefs, sleep quality, attitudes concerning the virus, the adherence to the measures, believing processes, and coping strategies/resilience patterns referring to COVID-19 in different study centers.

DETAILED DESCRIPTION:
A novel corona virus (SARS-CoV-2) has been identified as the cause of an outbreak of respiratory illness (corona virus disease COVID-19) all over the world. The COVID-19 pandemic is a public health emergency of international concern and poses a challenge to psychological resilience.

Studies reviewed the psychological impact of quarantine and reported negative psychological effects including post-traumatic stress symptoms, confusion, and anger, infection fears, frustration, boredom, inadequate supplies, inadequate information, financial loss, and stigma. A loss of daily structure and reduced social contacts were associated with frustration, boredom, reduced psychological-well being and psychological distress.

A recently conducted online questionnaire survey, investigating emotional responses and coping strategies of nurses, found sex differences in anxiety and fear referred to COVID-19 (women showed more severe anxiety and fear than men) and differences between participants from cities showing more anxiety and fear compared with participants from rural showing more sadness. The closer COVID-19 was to the participants, the stronger the anxiety and anger.

All these investigated psychological variables (i.e. anxiety, depression, boredom, loss of daily structure) have been found to impact the course and outcome of psychiatric disorders. Nowadays, COVID-19 is a pressure source with great influence, both for individuals and for the social public groups. Different individuals and groups may experience different levels of psychological crisis and patients with psychiatric disorders may experience more or less psychological symptoms than healthy control persons. According to a recent study, lithium, widely used to treat bipolar disorder, has been shown to exhibit antiviral activity and appears as a possible candidate for therapy of COVID-19. However, more research data are needed to develop evidence-driven strategies to reduce adverse psychological impacts and psychiatric symptoms during the pandemic.

Scientific questions

1. How do psychiatric patients experience the COVID-19 outbreak including quarantine and are there associations with affective symptoms and psychological distress? Is there a change in symptomatology during time? Are there differences to healthy controls, and between individuals with different diagnosis?
2. Is there a difference between psychiatric patients and healthy controls in regard to emotional response, cognition and behaviour during the COVID-19 pandemic and quarantine? Is there a difference between different psychiatric diagnosis groups?
3. Is there an association between consequences of social distance on lifestyle factors (nutrition, sleep quality, physical activity, substance abuse) and are there associations with psychological well-being/psychological symptoms in individuals with psychiatric disorder and controls? Is there a difference between different psychiatric diagnosis groups and healthy controls?
4. What do individuals with psychiatric disorders think about the COVID-19 related measures und quarantine regulations and how is the adherence to the measures? Are there associations between adherence and attitude towards COVID-19 measures? Is there a difference between patients and healthy controls? Is there a difference between different psychiatric diagnosis groups?
5. Are there sex and age differences in the investigated variables? (emotional response to COVID-19 outbreak, attitude towards measures, adherence)?
6. Is there a relationship between an infection with SARS-CoV-2 and disease course in psychiatric disorder? Is there a difference between different psychiatric diagnosis groups and healthy controls? Which role plays lithium treatment (prescribed beyond the study) in this context? The investigators hypothesize, loss of daily structure, reduced social contacts, loneliness, reduced psychiatric care, and other possible lifestyle changes due to the quarantine and social distancing measures, have a negative effect on psychological symptoms (depression, anxiety, somatisation, sleep quality) in individuals with psychiatric disorder compared to healthy controls. In contrast, resilience and positive cognition processes might be positively correlated to psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* voluntary participation

Exclusion Criteria:

* Subject refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on previous experience of the researchers working within the sector, we anticipated that it would be possible to recruit a conservative average of 100 psychiatric patients per outpatient clinic Thus, we aim to recruit at least 500 patients and 500 healthy controls in total which would be a large enough sample to conduct most subgroup analyses. Nevertheless, in case we can recruit a larger number of participants allowing further subgroup analysis it would be useful. The assumed response rate is 70 %.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Global symptom load (Anxiety, Somatisation, Depression, Global Symptom Index) | 1 year
  Brief Symptom Inventory-18 with higher scores meaning a worse outcome (more depression, anxiety and somatization); Each item is weighted on a 0-4 interval scale; Minimum = 0, Maximum = 72)
Depressive symptoms | 1 year
  Beck Depression Inventory-II with higher scores mean a worse Outcome (more depressive Symptoms; each item is weighted on a 0-3 interval scale; Minimum = 0, Maximum = 63)
Sleep disorders and Sleep Quality | 1 year
  Pittsburgh Sleep Quality Index (PSQI) with higher scores mean a worse Outcome (more sleeping disturbances; Each item is weighted on a 0-3 interval scale; Minimum = 0, Maximum = 63)

SECONDARY OUTCOMES:
Life style changes | 1 year
  Lifestyle Questions including physical activity, eating behavior, substance use, smoking
Food Craving | 1 year
  Food Craving Inventory (FCI) with higher scores mean a worse Outcome (more Food craving; Each item is weighted on a 0-4 interval scale; Minimum = 0, Maximum = 112)
COVID-19 associated fears and emotional responses to the pandemic | 1 year
  COVID-19 questionnaire with higher scores meaning a worse Outcome (more fears and negative emotions; each item is weighted on a 0-10 interval scale)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Reininghaus, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Department of Psychiatry and Psychotherapeutic Medicine, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided